CLINICAL TRIAL: NCT04426110
Title: Effect of Music Therapy in Pain and Anxiety Management for Patients Treated With Stitches in Emergency Department
Brief Title: Effect of Music Therapy in Pain and Anxiety Management for Patients Treated With Stitches
Acronym: PLAY
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200330
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Wound
Keywords: Wound; Stitches; Pain; Anxiety; Music
MeSH Terms: conditions — Wounds and Injuries; Pain; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Period 1 "Control": No Music. Wound stitches procedure conducted according to clinical practice.
- Period 2 "Music": Music by headphones. Wound stitches procedure conducted according to clinical practice

SUMMARY:
The aim of this study is to measure the effect of music therapy on pain and anxiety levels during stitches procedure in an adult emergency department.

DETAILED DESCRIPTION:
Wounds represent a frequent reason for admission to emergency department (5 to 7% of visits), inducing pain and anxiety due to the trauma itself and also to the treatment, stitches being the most frequently used procedure.

Alternative, non-pharmacologic strategies may help reduce pain and anxiety associated with painful bedside procedures. Music is one of them, easy to use and without any side effects.

Music therapy has already been shown to reduce pain and anxiety levels in children during medical procedures (blood test, vaccination, lumbar puncture) and in adults during surgical or anaesthetic procedures.

Our objective is to apply this technic to adults in emergency departments during stitches wound management.

This is a study before / after the implementation of a music therapy protocol during stiches wound management. During the music period, the participant will choose and listen to one of the five playlists (vocal jazz, instrumental jazz, piano, world music, Mozart) created by a professional music therapist, via headphones. There will be no change in stitches wound management.

Pain and anxiety levels will be measured by visual analog scale before, during and after the stitches procedure.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Acute skin wound with need for stitches
* National health service coverage
* No opposition

Exclusion Criteria:

* Conditions interfering with consent or measures (no French-fluent, acute intoxication, neurologic or psychiatric pathology)
* Wound requiring surgical exploration
* Wound localized on or around an ear
* Major insufficiency of auditory function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients visiting the emergency department for an acute skin wound with need for stitches.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Maximal pain level | Day 0
  Maximum pain level experienced during the procedure, measured by visual analog scale immediately after the procedure.

SECONDARY OUTCOMES:
Maximal anxiety level | Day 0
  Maximum anxiety level experienced during the procedure, measured by visual analog scale immediately after the procedure.
Final pain level | Day 0
  Final pain level measured by visual analog scale immediately after the procedure.
Final anxiety level | Day 0
  Final anxiety level measured by visual analog scale immediately after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Clément THIEBAUD, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Emergency Department Saint Antoine Hospital (AP-HP), Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cepeda MS, Carr DB, Lau J, Alvarez H. Music for pain relief. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD004843. doi: 10.1002/14651858.CD004843.pub2. PMID 16625614
- [Background] Klassen JA, Liang Y, Tjosvold L, Klassen TP, Hartling L. Music for pain and anxiety in children undergoing medical procedures: a systematic review of randomized controlled trials. Ambul Pediatr. 2008 Mar-Apr;8(2):117-28. doi: 10.1016/j.ambp.2007.12.005. PMID 18355741
- [Background] Kuhlmann AYR, de Rooij A, Kroese LF, van Dijk M, Hunink MGM, Jeekel J. Meta-analysis evaluating music interventions for anxiety and pain in surgery. Br J Surg. 2018 Jun;105(7):773-783. doi: 10.1002/bjs.10853. Epub 2018 Apr 17. PMID 29665028